CLINICAL TRIAL: NCT01184911
Title: Assessment of the Efficacy of Sulphadoxine-Pyrimethamine for Intermittent Preventive Treatment of Malaria in Pregnancy in Uganda
Brief Title: Sulphadoxine-Pyrimethamine for Intermittent Preventive Treatment of Malaria in Pregnancy in Uganda
Acronym: SP IPTp
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Research plan changed; no longer conducting clinical trial.
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Uganda Malaria Surveillance Project (Other)
Responsible Party: Grant Dorsey, University of California San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC5972
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Intermittent Preventive Treatment; Placental Malaria
Keywords: Malaria; Pregnancy
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SP (Experimental): Asymptomatic parasitemic pregnant women who receive the standard dose of sulfadoxine-pyrimethamine for prevention of placental malaria
  Interventions: Drug: Sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine — Sulfadoxine-pyrimethamine tablets, once
  Other Names: Kamsidar, Fansidar

SUMMARY:
The effectiveness of sulfadoxine-pyrimethamine (SP) as intermittent preventive treatment in pregnancy in malaria-endemic areas the effectiveness and efficacy of SP may be compromised by increased SP resistance. This study will evaluate the efficacy of SP by giving SP to asymptomatic parasitemic pregnant women and following them to determine the rates of parasite clearance.

ELIGIBILITY:
Inclusion Criteria:

* 16-26 weeks gestation based on LMP or ultrasound or fundal height
* Axillary temperature <37.5 degrees C
* Informed consent
* HIV status known and negative
* Blood smear positive for falciparum malaria

Exclusion Criteria:

* History of hypersensitivity reaction to SP or components of SP
* Axillary temperature ≥37.5 degrees C
* History of receipt of antimalarials or antibiotics with antimalarial activity* in the past month
* Residence > 30 km from the ANC clinic or unwillingness to return for follow-up visits
* Hemoglobin level < 5 gm/dL

  * These medications include all antimalarials, rifampin, doxycycline, clindamycin, tetracycline, erythromycin, azithromycin, chloramphenicol.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Parasite clearance | 42 days
  Clearance of parasites in pregnant women with asymptomatic parasitemia after administration of SP

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Ades, MD, MPH, Principal Investigator — University of California, San Francisco; Scott Filler, MD, DTM&H, Principal Investigator — Centers for Disease Control and Prevention; Moses Kamya, MBChB, MMed, MPH, PhD, Principal Investigator — Uganda Malaria Surveillance Project
Locations (1):
- Infectious Disease Research Center, Tororo, Tororo, Uganda

REFERENCES:
- See also: UMSP website — http://www.muucsf.org/umsp/about_umsp.html